CLINICAL TRIAL: NCT02038127
Title: Prospective Registry for Patients Undergoing Coronary Angiography and Percutaneous Coronary Intervention in Gangwon Province
Brief Title: Gangwon PCI Prospective Registry
Acronym: GWPCI
Status: Recruiting | Type: Observational
Sponsor: Yonsei University (Other)
Collaborators: Gangwon Cardiovascular Health Research Institute (Other)
Responsible Party: Principal Investigator, Young Jin Youn, MD, PhD, Assistant Professor, Yonsei University
Other Study IDs: GangwonPCI
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — CBC, Electrolyte, Chemistry, Cardiac biomarker, Platelet function test
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Comparison of

* Biolimus-eluting stent, Biomatrix, or Biomatrix Flex stent, Biosensors, Singapore
* Everolimus-eluting stent, Xience V, or Xience Prime, or Xience Xpedition stent, Abbott, USA
* Zotarolimus-eluting stent, Endeavor Resolute, or Endeavor Resolute Integrity stent Medtronic, USA in patients with coronary artery disease treated with percutaneous coronary intervention

ELIGIBILITY:
Inclusion Criteria:

* Age > 19 years
* Subject is able to verbally confirm understanding of risks, benefits and treatment alternatives of receiving the drug-eluting stent(s) and he/she or his/her legally authorized representative provides written informed consent prior to any study related procedure
* Subject must have significant stenosis (>50% by visual estimate) on a native or in-stent coronary artery
* Subject must have evidence of myocardial ischemia (e.g., stable, unstable angina, recent infarction, acute myocardial infarction, positive functional study or a reversible changes in the ECG consistent with ischemia). In subjects with coronary artery stenosis >75%, evidence of myocardial ischemia does not have to be documented

Exclusion Criteria:

* Subject has a known hypersensitivity or contraindication to any of the following medications: heparin, aspirin, clopidogrel, prasugrel, ticagrelor, biolimus A9, everolimus, zotarolimus, stainless steel, cobalt chromium, contrast media (Patients with documented sensitivity to contrast media, which can be effectively premedicated with steroid and diphenhydramine may be enrolled. However, those with true anaphylaxis to prior contrast media should not be enrolled.)
* Subject in use of systemic (intravenous) biolimus A9, everolimus or zotarolimus within 12 months.
* Female subject of childbearing potential, unless a recent pregnancy test is negative, who possibly plans to become pregnant any time after enrollment into this study
* Subject planned an elective surgical procedure that would necessitate interruption of antiplatelet during the first 12 months post enrollment
* Subject with non-cardiac co-morbid condition with life expectancy < 2 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* Subject with cardiogenic shock at presentation
* Subject who are actively participating in another drug or device investigational study, who have not completed the primary end point follow-up period

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were at least 18 years of age, who have stable coronary artery disease (CAD) or acute coronary syndrome (ACS), including myocardial infarction (MI) with or without ST-segment elevation will be included in the study.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2013-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Device-oriented composite outcome | 24 months
  Device-oriented composite consisted of cardiac death, MI not clearly attributable to a nontarget vessel, and clinically indicated TLR at 24-month clinical follow-up

SECONDARY OUTCOMES:
Patient-oriented composite outcome | 24 months
  Patient-oriented composite consisted of all-cause mortality, any MI, and any revascularization at 24-month clinical follow-up
Target vessel revascularization | 12 months
Target vessel revascularization | 24 months
ARC defined stent thrombosis | 12 months
ARC defined stent thrombosis | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Junghan Yoon, M.D., Ph.D., Principal Investigator — Yonsei University
Locations (3):
- South Korea (3):
  - Chuncheon Hallym University Hospital, Chuncheon, Gangwon-do
  - Yonsei University Wonju Christian Hospital, Wŏnju, Gangwon-do
  - Korea University Guro Hospital, Seoul

REFERENCES:
- [Derived] Jeon HS, Youn YJ, Lee JH, Park YJ, Son JW, Lee JW, Ahn MS, Ahn SG, Kim JY, Yoo BS, Yoon J. Safety and Efficacy of Two Ultrathin Biodegradable Polymer Sirolimus-Eluting Stents in Real-World Practice: Genoss DES Stents Versus Orsiro Stents From a Prospective Registry. Clin Cardiol. 2024 Dec;47(12):e70060. doi: 10.1002/clc.70060. PMID 39691038
- [Derived] Jeon HS, Kim YI, Lee JH, Park YJ, Son JW, Lee JW, Youn YJ, Ahn MS, Kim JY, Yoo BS, Ko SM, Ahn SG. Failed Thrombus Aspiration and Reduced Myocardial Perfusion in Patients With STEMI and Large Thrombus Burden. JACC Cardiovasc Interv. 2024 Oct 14;17(19):2216-2225. doi: 10.1016/j.jcin.2024.07.016. Epub 2024 Sep 18. PMID 39297854
- [Derived] Youn YJ, Jeon HS, Kim YI, Lee JH, Park YJ, Cho DH, Son JW, Lee JW, Ahn MS, Ahn SG, Kim JY, Yoo BS, Lee SH, Yoon J. Impact of the ultra-long 48 mm drug-eluting stent on procedural and clinical outcomes in patients with diffuse long coronary artery disease. Clin Cardiol. 2023 Apr;46(4):416-424. doi: 10.1002/clc.23997. Epub 2023 Feb 20. PMID 36807273